CLINICAL TRIAL: NCT01427504
Title: A Bioequivalence Study to Evaluate the Potential for Drug-drug Interactions Between Boceprevir 800mg Thrice Daily and the HIV Non-nucleoside Reverse Transcriptase Inhibitor Etravirine 200mg Twice Daily in HIV/(Hepatitis C Virus) (HCV) Negative Volunteers
Brief Title: Potential for Drug-drug Interactions Between Boceprevir and Etravirine in HIV/Hepatitis C Virus Negative Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 11-1046
Record Dates: First submitted 2011-08-24; First posted 2011-09-01 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis C; HIV
Keywords: HCV; HIV
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1a (Experimental): Sequence 1,2,3: boceprevir only, then etravirine only, then both boceprevir and etravirine.
  Interventions: Drug: boceprevir; etravirine
- Sequence 1b (Experimental): Sequence 1,3,2: boceprevir only, then both boceprevir and etravirine, then etravirine only.
  Interventions: Drug: boceprevir; etravirine
- Sequence 2a (Experimental): Sequence 2,1,3: etravirine only, then boceprevir only, then both boceprevir and etravirine.
  Interventions: Drug: boceprevir; etravirine
- Sequence 2b (Experimental): Sequence 2,3,1: etravirine only, then both boceprevir and etravirine, then boceprevir only.
  Interventions: Drug: boceprevir; etravirine
- Sequence 3a (Experimental): Sequence 3,1,2: both boceprevir and etravirine, then boceprevir only, then etravirine only.
  Interventions: Drug: boceprevir; etravirine
- Sequence 3b (Experimental): Sequence 3,2,1: Both boceprevir and etravirine, then etravirine only, then boceprevir only.
  Interventions: Drug: boceprevir; etravirine

INTERVENTIONS:
Drug: boceprevir; etravirine — boceprevir tablets 800 mg, every 8 hours x 11-14 days. etravirine tablets 200 mg, every 12 hours x 11-14 days.

SUMMARY:
The investigators believe that boceprevir's drug concentrations will be reduced when administered in combination with etravirine. The investigators believe that etravirine's drug concentrations will be increased when administered in combination with boceprevir. Additionally, the investigators believe that boceprevir and etravirine are safe when administered alone or in combination.

DETAILED DESCRIPTION:
To investigate the potential for drug interactions between boceprevir and etravirine, participants will receive each drug alone and the drugs in combination for 11-14 days. The pharmacokinetics of boceprevir and etravirine when given in combination vs. alone will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-60 years
* Absence of HIV-1 and HCV antibodies at screening
* Ability and willingness to give written informed consent before the first trial-related activity

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Active alcohol or drug abuse that, in the opinion of the investigators, would interfere with adherence to study requirements.
* Participation in any investigation drug study within 30 days prior to study.
* Currently active or chronic gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease or malignancy requiring pharmacologic treatment, and/or if in the opinion of the investigator, would affect study participation, safety, or integrity of results.
* Use of concomitant medication, including investigational, prescription, and over-the-counter products and dietary supplements with the following exceptions:aspirin, acetaminophen, once daily multivitamins, mineral supplements and hormonal oral contraceptives (other than those that contain drospirenone). Concomitant medications other than those listed above must have been discontinued at least 14 days before study entry.
* Currently active dermatitis or urticaria or diagnosis of eczema or psoriasis.
* History of significant drug allergy (i.e., anaphylaxis and/or angioedema)
* Subjects with the following laboratory abnormalities at screening as defined by the 2004 Division of AIDS Table for grading the Severity of Adult and Pediatric Adverse Events and in accordance with the normal ranges of the trial clinical laboratory: serum creatinine grade 1 or greater (>1.1 x upper limit of laboratory normal range (ULN); hemoglobin grade 1 or greater (≤ 10.9 g/dL); platelet count grade 1 or greater (≤ 124.999 x 109/L); absolute neutrophil count grade 1 or greater (≤ 1.3 x 109/L); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) grade 1 or greater (≥ 1.25 x ULN); total bilirubin grade 1 or greater (≥ 1.1 x ULN), any other laboratory abnormality of grade 2 or above

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kiser, PharmD, Principal Investigator — Univesity of Colorado Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured at the University of Colorado Hospital beginning September 1, 2011 and ended on October 4, 2011.
Pre-assignment Details: There were 8 subjects that were excluded from trial before assignment to groups; 5 due to personal reasons, 2 due to elevated bilirubin, and 1 due to elevated serum creatinine.
Groups:
- Sequence 1a: Sequence 1,2,3: boceprevir 800 mg three times daily alone, then etravirine 200 mg twice daily only, then both boceprevir 800 mg three times daily and etravirine 200 mg twice daily were each given for 11-14 days. Each intervention was followed by a 14 day washout period before the next sequence was started.
- Sequence 1b: Sequence 1,3,2: boceprevir 800 mg three times daily alone, then etravirine 200 mg twice daily only, then both boceprevir 800 mg three times daily and etravirine 200 mg twice daily were each given for 11-14 days. Each intervention was followed by a 14 day washout period before the next sequence was started.
- Sequence 2a: Sequence 2,1,3: boceprevir 800 mg three times daily alone, then etravirine 200 mg twice daily only, then both boceprevir 800 mg three times daily and etravirine 200 mg twice daily were each given for 11-14 days. Each intervention was followed by a 14 day washout period before the next sequence was started.
- Sequence 2b: Sequence 2,3,1: boceprevir 800 mg three times daily alone, then etravirine 200 mg twice daily only, then both boceprevir 800 mg three times daily and etravirine 200 mg twice daily were each given for 11-14 days. Each intervention was followed by a 14 day washout period before the next sequence was started.
- Sequence 3a: Sequence 3,1,2: boceprevir 800 mg three times daily alone, then etravirine 200 mg twice daily only, then both boceprevir 800 mg three times daily and etravirine 200 mg twice daily were each given for 11-14 days. Each intervention was followed by a 14 day washout period before the next sequence was started.
- Sequence 3b: Sequence 3,2,1: boceprevir 800 mg three times daily alone, then etravirine 200 mg twice daily only, then both boceprevir 800 mg three times daily and etravirine 200 mg twice daily were each given for 11-14 days. Each intervention was followed by a 14 day washout period before the next sequence was started.
Period: Overall Study
Arm/Group | Sequence 1a | Sequence 1b | Sequence 2a | Sequence 2b | Sequence 3a | Sequence 3b
Started | 4 | 3 | 4 | 6 | 3 | 6
Received Boceprevir | 4 | 3 | 3 | 5 | 2 | 4
Received Etravirine | 4 | 2 | 4 | 6 | 2 | 4
Received Combination | 4 | 3 | 3 | 6 | 3 | 6
Completed | 4 | 2 | 3 | 5 | 2 | 4
Not Completed | 0 | 1 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1a | Sequence 1b | Sequence 2a | Sequence 2b | Sequence 3a | Sequence 3b | Total
Number analyzed (Participants) | 4 | 3 | 4 | 6 | 3 | 6 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 4 | 3 | 3 | 6 | 3 | 6 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.4) | 35.6 (8.0) | 33.3 (9.8) | 25.9 (3.8) | 42.7 (16.8) | 32.4 (9.3) | 34.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3 | 2 | 6 | 14
  Male | 3 | 1 | 4 | 3 | 1 | 0 | 12
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 6 | 3 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Boceprevir AUC Pharmacokinetics
Description: Determine boceprevir area-under-the concentration time curve (AUC) when administered alone.
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, and 8 hours post dose on day 11-14
Population: The number of participants was based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Boceprevir AUC: Geometric mean of boceprevir AUC administered alone.
Arm/Group | Boceprevir AUC
Number analyzed (Participants) | 20
ng*hr/mL | 4601 (47)

2. Primary Outcome: Boceprevir Cmax Pharmacokinetics
Description: Determine the Cmax of boceprevir when administered alone.
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, and 8 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Boceprevir Cmax: Geometric mean of boceprevir Cmax when administered alone.
Arm/Group | Boceprevir Cmax
Number analyzed (Participants) | 20
ng/mL | 1423 (43) [0.66 to 0.91]

3. Primary Outcome: Boceprevir C8 Pharmacokinetics
Description: Determine boceprevir 8 hour concentration when administered alone.
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, and 8 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Boceprevir C8: Geometric mean of boceprevir Cmax when administered alone.
Arm/Group | Boceprevir C8
Number analyzed (Participants) | 20
ng/mL | 106 (64)

4. Primary Outcome: Etravirine AUC Pharmacokinetics
Description: Determine etravirine area under the concentration vs. time curve (AUC)when administered alone.
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Etravirine AUC: Geometric mean of etravirine AUC when administered alone.
Arm/Group | Etravirine AUC
Number analyzed (Participants) | 20
ng*hr/mL | 7698 (33)

5. Primary Outcome: Etravirine Cmax Pharmacokinetics
Description: Determine etravirine Cmax when administered alone
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Etravirine Cmax: Geometric mean of etravirine Cmax when administered alone.
Arm/Group | Etravirine Cmax
Number analyzed (Participants) | 20
ng/mL | 900 (29)

6. Primary Outcome: Etravirine Cmin Pharmacokinetics
Description: Determine etravirine Cmin when administered alone
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Etravirine Cmin: Geometric mean of etravirine Cmin when administered alone.
Arm/Group | Etravirine Cmin
Number analyzed (Participants) | 20
ng/mL | 439 (46)

7. Primary Outcome: Boceprevir AUC Pharmacokinetics Coadministered With Etravirine
Description: Determine boceprevir AUC when coadministered with etravirine. [Ratio = boceprevir administered with etravirine/ boceprevir alone]
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, and 8 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Boceprevir AUC Coadministered With Etravirine: Geometric mean ratio of boceprevir AUC when coadministered with etravirine
Arm/Group | Boceprevir AUC Coadministered With Etravirine
Number analyzed (Participants) | 20
Ratio | 1.10 [0.94 to 1.28]

8. Primary Outcome: Boceprevir Cmax Pharmacokinetics Coadministered With Etravirine
Description: Determine boceprevir Cmax when coadministered with etravirine. [Ratio = boceprevir administered with etravirine / boceprevir alone]
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, and 8 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Boceprevir Cmax Coadministered With Etravirine: Geometric mean ratio of boceprevir Cmax when coadministered with etravirine
Arm/Group | Boceprevir Cmax Coadministered With Etravirine
Number analyzed (Participants) | 20
Ratio | 1.10 [0.94 to 1.29]

9. Primary Outcome: Boceprevir C8 Pharmacokinetics Coadministered With Etravirine
Description: Determine boceprevir 8 hour concentration when coadministered with etravirine. [Ratio = boceprevir administered with etravirine / boceprevir administered alone]
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, and 8 hours post dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Boceprevir C8 Coadministered With Etravirine: Geometric mean ratio of boceprevir C8 when coadministered with etravirine
Arm/Group | Boceprevir C8 Coadministered With Etravirine
Number analyzed (Participants) | 20
Ratio | 0.88 [0.66 to 1.17]

10. Primary Outcome: Etravirine AUC Pharmacokinetics Coadministered With Boceprevir
Description: Determine etravirine AUC when coadministered with boceprevir. [Ratio = Etravirine administered with bocepreivr / etravirine administered alone]
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours Post-dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Etravirine AUC Coadministered With Boceprevir: Geometric mean ratio of etravirine AUC when coadministered with boceprevir
Arm/Group | Etravirine AUC Coadministered With Boceprevir
Number analyzed (Participants) | 20
Ratio | 0.77 [0.66 to 0.91]

11. Primary Outcome: Etravirine Cmax Pharmacokinetics Coadministered With Boceprevir
Description: Determine etravirine Cmax when coadministered with boceprevir. [Ratio = etravirine administered with boceprevir / etravirine administered alone]
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Etravirine Cmax: Geometric mean ratio of etravirine Cmax when coadministered with boceprevir
Arm/Group | Etravirine Cmax
Number analyzed (Participants) | 20
Ratio | 0.76 [0.68 to 0.85]

12. Primary Outcome: Etravirine Cmin Pharmacokinetics Coadministered With Boceprevir
Description: Determine etravirine Cmin when coadministered with boceprevir. [Ratio = etravirine administered with boceprevir / etravirine administered alone]
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose on day 11-14
Population: The number of participants is based on the number of subjects that completed all three sequences of medication.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Etravirine Cmin Coadministered With Boceprevir: Geometric mean ratio of etravirine Cmin when coadministered with boceprevir
Arm/Group | Etravirine Cmin Coadministered With Boceprevir
Number analyzed (Participants) | 20
Ratio | 0.71 [0.54 to 0.95]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Adverse events were verbally assessed by study investigators. Laboratory tests were performed at baseline and at all three intensive pharmacokinetic study visits. Clinical and laboratory adverse events were graded using the 2004 Division of AIDS table for grading the severity of adult and pediatric adverse experiences.
Groups:
- Boceprevir Alone: Subjects took boceprevir alone, 800 mg thrice daily, for 10-14 days.
- Etravirine Alone: Subjects took etravirine alone, 200 mg twice daily, for 10-14 days
- Boceprevir Coadministered With Etravirine: Boceprevir, 800 mg thrice daily, coadministered with etravirine, 200 mg twice daily for 10-14 days.
Arm/Group | Boceprevir Alone | Etravirine Alone | Boceprevir Coadministered With Etravirine
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/22 | 5/25
Other Adverse Events (participants affected / at risk) | 19/21 | 11/22 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir Alone (N=21) | Etravirine Alone (N=22) | Boceprevir Coadministered With Etravirine (N=25)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Increased energy, anxiety, nervousness, insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presumed Viral Illness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boceprevir Alone (N=21) | Etravirine Alone (N=22) | Boceprevir Coadministered With Etravirine (N=25)
Altered Taste (Gastrointestinal disorders) | 18 (18) | 0 (0) | 16 (16)
Headache (General disorders) | 4 (4) | 5 (5) | 4 (4)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3)
Hypokalemia (General disorders) | 4 (4) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 4 (4)

LIMITATIONS AND CAVEATS:
1. Healthy volunteer study does not take into account other medications being prescribed to treat the co-infected population.
2. An interaction at the level of enzyme induction is difficult to rule out since we sampled etravirine over 12 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No